CLINICAL TRIAL: NCT05363631
Title: Phase I/II Study of Seleno-L Methionine (SLM) in Sequential Combination With Fixed Doses and Schedules of Axitinib and Pembrolizumab (SAP) in Locally Advanced and Metastatic Clear Cell Renal Cell Carcinoma (ccRCC)
Brief Title: Seleno-L Methionine (SLM)-Axitinib-Pembrolizumab
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mohammed Milhem (Other)
Collaborators: University of Iowa (Other)
Responsible Party: Sponsor-Investigator, Mohammed Milhem, Clinical Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202104398
Record Dates: First submitted 2022-05-02; First posted 2022-05-06 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Clear Cell Renal Cell Carcinoma; Clear Cell Renal Cell Carcinoma Metastatic
MeSH Terms: conditions — Carcinoma, Renal Cell; Clear-cell metastatic renal cell carcinoma | interventions — Selenomethionine; Axitinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Seleno-L Methionine (SLM) in Combination with Axitinib and Pembrolizumab (Experimental): SLM only will be taken by mouth during a two-week run in period. Then patients will receive SLM and Axitinib drugs by mouth, and Pembrolizumab intravenously (IV), at the start of each 21 day cycle.
  Interventions: Drug: Selenomethionine (SLM); Drug: Axitinib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Selenomethionine (SLM) — Selenium (Se) is a natural element present in the earth's crust often in association with sulfur-containing compounds. Humans get their dietary requirements mainly from food. In this study Selenium will be administered in the chemical composition of selenomethionine (SLM)
Drug: Axitinib — Axitinib is a small molecule tyrosine kinase inhibitor.
Drug: Pembrolizumab — Pembrolizumab is a type of immunotherapy

SUMMARY:
The purpose of this research study is to test the safety and effectiveness of Seleno-L Methionine (SLM) when combined with the standard dose and schedule of Axitinib and Pembrolizumab in patients who have locally advanced or metastatic clear cell renal cell carcinoma (ccRCC).

DETAILED DESCRIPTION:
The proposed study is a single arm, open-label Phase I/II trial of Seleno-L Methionine (SLM) in sequential combination with the standard dose and schedule of Axitinib and Pembrolizumab in previously untreated patients with advanced ccRCC. The hypothesis is that adding SLM to the Pembrolizumab and Axitinib combination will improve efficacy without added toxicity.

This is a two-part study:

* Escalation Part 1: The study will begin with a dose-escalation study to find the maximum tolerated dose (MTD) of study drug, SLM.
* Expansion Part 2: Once the appropriate dose of SLM is determined, the second part of the study will begin.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, an individual must meet all the following criteria:

* Written and voluntary informed consent.
* Histologically and radiologically confirmed locally advanced or metastatic ccRCC. Locally advanced is defined as non resectable in the opinion of the treating providers. Participants must be treatment naïve in metastatic setting. Prior immunotherapy treatment in adjuvant setting is allowed.
* > 18 years of age
* At least one Response Evaluation Criteria in Solid Tumors (RECIST 1.1)-defined target lesion that has not been irradiated
* Eastern Cooperative Oncology Group performance status of 0 (fully active, able to carry on all pre-disease performance without restriction) or 1 (restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, such as light housework or office work).
* Renal function (creatinine level within normal institutional limit, or creatinine clearance >15 mL/min/1.73 m2 for patients with creatinine levels above institutional normal, calculated using the Cockcroft-Gault formula).
* Liver function (AST/ALT <3.0 X institutional upper limit of normal OR < 5 x institutional upper limit of normal in cases of liver metastases; Total bilirubin ≤ 1.5 times ULN.)
* Adequate hematological lab values including

  * Absolute Neutrophil Count (ANC) ≥ 1.0 x 109/L
  * Platelets ≥ 100 x 109/L
  * Hemoglobin ≥ 7.0 g/dL
* Has adequately controlled BP with or without antihypertensive medications, defined as BP ≤150/90 mm Hg with no change in antihypertensive medications within 1 week before randomization/allocation.
* Female subjects of childbearing potential and non-sterilized male subjects who intend to be sexually active during the study must agree to use a highly effective method of contraception from the time of screening, throughout the total duration of the drug treatment, and during the 6 month post-drug washout period. See section 5.6 for full details.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Patients with a prior or concurrent malignancy whose natural history or treatment may have the potential to interfere with the safety or efficacy assessment of the investigational regimen.
* Untreated metastases in the central nervous system.
* Pregnant or breastfeeding.
* Present use or anticipated need for cytochrome P450 (CYP) 3A4-inhibiting, CYP3A4-inducing drugs (e.g., ketoconazole, itraconazole, clarithromycin, atazanavir, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, and voriconazole, rifampin, phenytoin, carbamazepine, rifabutin, rifapentine, phenobarbital, and St. John's wort, bosentan, efavirenz, etravirine, modafinil, and nafcillin).
* Myocardial infarction, uncontrolled angina, congestive heart failure, or cerebrovascular accident within previous 6 months. Participants with history of deep vein thrombosis or pulmonary embolism, at provider discretion.
* Major surgery within 4 weeks of starting study treatment.
* Patients with HIV infection with CD4+ T-cell (CD4+) counts < 350 cells/uL
* Patients with HIV infection and a history of AIDS-defining opportunistic infections

No exclusions will be made based on sex, race, or ethnic background.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2022-09-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase I - Dose limiting toxicities using National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.0 | From the initiation of treatment through three years
  To examine the toxicity related to the therapy by measuring the number of treatment related adverse events in patients
Phase II - Objective Response Rate (ORR) | From the initiation of treatment through three years
  ORR will be defined as the proportion of patients with a best overall response of complete response (CR) or partial response (PR) per RECIST v1.1

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From the initiation of treatment through three years
  PFS will be defined as the time from treatment initiation to the date of first documentation of disease progression or death due to any cause
Overall survival (OS) | From the initiation of treatment through three years
  OS will be defined as the time from treatment initiation to the date of death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Milhem, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No